CLINICAL TRIAL: NCT06605976
Title: Evaluating the Impact of Ambient AI on Documentation Efficiency and Clinician Burnout in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samaritan Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB23-072
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Burnout; Clinical Documentation Efficiency
Keywords: clinical documentation; burnout; scribe; ambient AI; DAX CoPilot; randomized control trial; electronic health record; acceptance and use of technology; patient satisfaction
MeSH Terms: conditions — Burnout, Psychological; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAX CoPilot Group (Experimental): Participants in this arm were given a DAX CoPilot license and asked to use it for clinical documentation in the EHR.
  Interventions: Behavioral: DAX CoPilot Group
- Control group (No Intervention): Participants in this arm were not given a DAX CoPilot license and were asked to use standard methods for clinical documentation in the EHR.

INTERVENTIONS:
Behavioral: DAX CoPilot Group — Participants in this group were given a license for DAX CoPilot and asked to use it for clinical documentation.
  Arms: DAX CoPilot Group

SUMMARY:
This clinical trial aims to evaluate the effectiveness of an ambient listening AI product, DAX CoPilot, in improving clinical documentation efficiency and reducing clinician burnout in primary care settings. Researchers will compare results from a group who was given a license to use DAX CoPilot to a group who was not given a license. Participants in the DAX group will use DAX CoPilot system for EHR documentation and participants in the control group will use use standard EHR documentation methods. Participants will also be asked to complete surveys and assessments related to their views on technology and experiences of burnout.

DETAILED DESCRIPTION:
This pilot study aims to evaluate the effectiveness of an ambient listening AI product in improving clinical documentation efficiency and patient satisfaction, reducing clinician burnout in primary care settings, and improving operational implementation strategies by harnessing end-user psychology. Employing a randomized, prospective design, the study involved 25 clinicians who were given an ambient listening AI product (DAX CoPilot) after a 1 month baseline period and asked to use it for clinical documentation with a focus on problem-focused visits over a 3-month period, with a control group of 20 clinicians continuing traditional documentation methods. The primary outcomes include changes in documentation efficiency (measured through metrics such as time spent on documentation per patient) and clinician burnout (assessed using the validated Mini-Z 2.0 burnout inventory). Secondary outcomes involve patient satisfaction with clinicians' use of the AI tool and examining end-user technology acceptance among clinicians using a survey based on the Unified Theory of Acceptance and Use of Technology (UTAUT). The study aims to provide insights into the potential of AI-assisted documentation tools in enhancing clinical workflow and addressing the growing concern of clinician burnout.

ELIGIBILITY:
Inclusion Criteria:

1. Licensed Clinicians: Independently licensed clinicians (MDs, DOs, NPs, PAs) who have been actively practicing at Samaritan Health Services for at least 6 months.
2. Primary Care Only: Providers must have a listed specialty of family medicine, internal medicine, or pediatrics, and currently practice primarily in a primary or urgent care clinic.
3. Provider has an Apple iPhone and is willing to install Epic Haiku.

Exclusion Criteria:

1. Inpatient-Only Clinicians: Exclude clinicians who only, or primarily, work in inpatient settings, as documentation needs and challenges may differ significantly from those in outpatient settings.
2. Trainees: Exclude medical students and residents due to their varying levels of experience and dependence on supervisory oversight.
3. Minimum Outpatient Encounters: Exclude clinicians with fewer than 100 outpatient encounters per month to focus on those with a significant workload in outpatient settings.
4. Android Smartphones Users: Clinicians may not use Android, or generally any non-Apple or non-iOS smartphones, given the software limitations of the selected intervention technology.
5. Corrective Action: Exclude clinicians facing dismissal, corrective, or disciplinary action.
6. Scheduled leave longer than 3 weeks during the study period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Documentation efficiency | From baseline to the end of the 3 month experimental period
  Compare average documentation, workload, and InBasket metrics (tracked by Epic Signal and through a custom data pull for SHS) before and after the implementation of ambient AI among the intervention and control groups; time in notes per appointment, time in notes per scheduled day, progress note length, note composition, time outside scheduled hours, time outside of 7 AM to 7 PM, pajama time, visits closed same day, time in InBasket per appointment, InBasket message turnaround time

SECONDARY OUTCOMES:
Burnout | From baseline to the end of the 3 month experimental period
  Clinician burnout as assessed using the Mini-Z 2.0 burnout inventory

OTHER OUTCOMES:
Patient satisfaction | 3 months experimental period
  Patient satisfaction with the experience of the clinician using DAX CoPilot via a patient survey after a visit in which it was used

CONTACTS AND LOCATIONS:
Locations (1):
- Samaritan Health Services, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided